CLINICAL TRIAL: NCT06047431
Title: A Phase Ⅰ Study to Evaluate the Pharmacokinetics, Safety, Tolerability and Efficacy of QL1706H in Advanced Solid Tumors
Brief Title: A Study of QL1706H in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QL1706H-101
Record Dates: First submitted 2023-07-03; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1706H (Experimental): Part 1 (Dose escalation): QL1706H will be administered in sequential cohorts each receiving 1 dose of QL1706H by subcutaneous injection on day 1 and QL1706 by IV infusion on day 22, from then on will recieve QL1706 on day 1 of every 21-day cycle (3 weeks). Dose escalation will continue until the projected cohorts has been finished.
  Part 2 (Dose Exploration): The PK parameters of QL1706H will be tested at different administration intervals.
  Interventions: Drug: QL1706H

INTERVENTIONS:
Drug: QL1706H — QL1706H is the subcutaneousely administered formulation of QL1706, it contains two unique monoclonal antibodies.

SUMMARY:
This is an open-label, Phase Ⅰ study of QL1706H in patients with advanced solid tumors. The study will evaluate the pharmacokenetics, safety, tolerability and preliminary efficacy of QL1706H.

DETAILED DESCRIPTION:
The study is composed of 2 parts. Part 1 is a dose-escalation study to explore the pharmacokenetics (PK), safety, and tolerability of QL1706H. Part 2 of the study will explore the PK characteristics of differente intervals and sites of administration. All the PK parameters will determine the recommended Phase 2 dose (RP2D).

The study was divided into screening/baseline, treatment and follow-up periods. Safety monitoring will be conducted throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects participate voluntarily and sign informed consent.
* Patients with Pathologically confirmed metastatic or recurrent malignant solid tumors, failure or intolerance of at least first-line treatment and unsuitable for radical treatment such as surgery
* Subject has at least one measurable lesion according to RECIST (V1.1) evaluation criteria.
* Eastern Cooperative Oncology Group (ECOG) score was 0 or 1.
* The extension of life is more than 3 months
* Vital organs' function is adequate for enrolling
* Subjects agree to use effective contraceptive measures.Women who have not been pregnant or breastfeeding.
* Before the first use of the investigational drug, all the reversible toxicity of the previous antitumor therapy returned to ≤1 (according to CTCAE V5.0),Excluding any grade of hair loss and pigmentation, grade 2 or less peripheral sensory neuropathy, and other abnormalities that the investigator and/or sponsor assessed to outweigh the risk of toxicity.

Exclusion Criteria:

* Active autoimmune diseases that exist within 2 years prior to the first use of the investigational drug and require systemic treatment.
* There are known past grade 3 or 4 immune-related adverse events associated with antitumor immunotherapy.
* Symptomatic central nervous system (CNS) metastasis, pia metastasis or spinal cord compression due to metastasis prior to signing informed consent.
* Subjects with any of the following cardiovascular diseases that seriously endanger the safety of the subjects or affect the completion of the study
* Subjects with diseases that are planned to be treated with systemic corticosteroids or other immunosuppressive drugs during the study period
* Prior treatment with cytotoxic T lymphocyte-associated antigen-4 (CTLA-4) inhibitor combined with programmed cell death protein-1 (PD-1) inhibitor, or CTLA-4 inhibitor combined with PD-L1 inhibitor.
* Had received chemotherapy, targeted therapy, biotherapy, endocrine therapy, immunotherapy and other anti-tumor treatments within 4 weeks before the first use of experimental drugs
* Subjects with positive antibodies to HIV;Treponema pallidum antibody positive;HBsAg positive patients with VIRAL DEoxy ribonucleic acid (HBV DNA) >2000 IU/ mL or 10^4 copy number/mL should receive antiviral therapy according to local treatment guidelines and be willing to receive antiviral therapy throughout the study period.Hepatitis C virus antibody positive and viral ribonucleic acid (HCV RNA) positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Minimum Serum Drug Concentration ( Ctrough) | one cycle (3 weeks)
  The minimum serum drug concentration and area under serum concentration-time curve after single administration of QL1706H.

SECONDARY OUTCOMES:
Safety and tolerability | one cycle (3 weeks)
  Safety and tolerability, as defined by the rate of treatment-related adverse events as assessed by NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Lu, Doctor, Principal Investigator — Tianjin Cancer Hospital

IPD SHARING:
Plan to Share IPD: No